CLINICAL TRIAL: NCT06273306
Title: Towards Telemonitoring in Immune-Mediated Inflammatory Diseases: Implementation of a Mixed Attention Model
Brief Title: Towards Telemonitoring in Immune-Mediated Inflammatory Diseases: Implementation of a Mixed Attention Model (IMIDOC)
Acronym: IMIDOC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HULP.PI-4519; PI22/00777 (Other Grant/Funding Number: Fondo de investigaciones sanitarias.Instituto de Salud Carlos III)
Record Dates: First submitted 2024-01-08; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-12

CONDITIONS: Telemedicine; Telehealth; eHealth; Rheumatic Diseases; Arthritis, Rheumatoid; Spondylarthritis
MeSH Terms: conditions — Rheumatic Diseases; Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital care (Experimental): User of mobile APP for telemonitoring
  Interventions: Device: IMIDOC
- Traditional care (No Intervention): Monitoring in face-to-face visits

INTERVENTIONS:
Device: IMIDOC — Patient´s Mobile App for recording clinical data
  Arms: Digital care

SUMMARY:
The main objective is to evaluate the implementation of a hybrid care model called the mixed attention model (MAM) in clinical practice and to evaluate whether its implementation improves clinical outcomes compared to conventional follow-up.

This is a multicenter prospective observational study involving 360 patients with rheumatoid arthritis (RA) and Spondylarthritis (SpA) from five Spanish Hospitals. Patients will be followed-up by the MAM protocol, which is a care model that incorporates the use of digital tool consisting of a mobile application (App) that patients can use at home and that professionals can review asynchronously to detect incidents and to follow their patients; clinical evolution between face-to-face visits. Another group of patients, whose follow-up will be conducted in accordance with a traditional face-to-face care model, will be assessed as the control group. Sociodemographic characteristics, treatments, laboratory parameters, assessment of tender and swollen joints, visual analogue scale for pain and electronic patient reported outcome reports (ePROs) will be collected for all subjects. In the MAM group, these items will be self-assessed both by the mobile App and during face-to-face visits with rheumatologist, who will do the same for patients included in the traditional care model. Patients will be able to report any incidence related to their disease or treatment through the mobile App.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with Rheumatoid Arthritis or Spondylarthritis
* Treatment with biologic or targeted disease modifying antirheumatic drugs.
* Ability to use smartphone.

Exclusion Criteria:

* only patients with conditions that hinder or prevent the use of a mobile application (blindness, mental retardation, dementia, digitalfilliteracy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the primary objective, composite endpoints that consider the viability, adherence and degree of satisfaction of the MAM are included | 24 months
  * Number of interactions in activity and electronic patient reported outcomes (ePRO) questionnaires per month.
  * Number of reported incidences per month.
  * Average time to contact the patient after reporting an incident.
  * Average number of interactions in educational material and other content per month.
  * Adherence to follow-up through the mixed atenttion model (MAM) will be evaluated through the number of visits and time per visit to the digital platform.
  * Percentage of incidents resolved telematically.
  * Average weekly hours that the digital clinician takes to review the professional's website and resolve incidents
  * Professionals and patients´ satisfaction will be assessed through the Net-Promoter-Score (NPS). Values from 0 to 6 ( detractors), 6-8 ( passives) and 9-10 promoters.

SECONDARY OUTCOMES:
To identify features associated with adherence to follow-up through the MAM. | 24 months
  * A 22-item self-administered survey adapted from the Unified Theory of Acceptance and Use of Technology (UTAUT) model will be used to measure app acceptance and intention to use: the variables will measured with 7-point scales for all model components as in the original UTAUT, where 1 equalled the negative end (fully disagree) and 7 the positive end of the scale (fully agree).
  * Agreement between patients' self-assessment and clinician assessment will be assessed comparing face-to-face visits at 6-months intervals with the closest assessment in the digital solution.
  * Number of face-to-face visits are avoided with the mixed atenttion model (MAM) in patients with stable disease activity.
  * Patients' eHealth literacy will be measured using the validated Spanish version of the eHealth Literacy Scale (eHEALS), measured on a 5-point scale in the range from 1 (strongly disagree) to 5 (strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Chamaida Plasencia-Rodríguez, PhD, Principal Investigator — Hospital Universitario La Paz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novella-Navarro M, Iniesta-Chamorro JM, Benavent D, Bachiller-Corral J, Calvo-Aranda E, Borrell H, Berbel-Arcobe L, Navarro-Compan V, Michelena X, Lojo-Oliveira L, Arroyo-Palomo J, Diaz-Almiron M, Garcia Garcia V, Monjo-Henry I, Gomez Gonzalez CM, Gomez EJ, Balsa A, Plasencia-Rodriguez C. Toward Telemonitoring in Immune-Mediated Inflammatory Diseases: Protocol for a Mixed Attention Model Study. JMIR Res Protoc. 2024 Apr 22;13:e55829. doi: 10.2196/55829. PMID 38501508